CLINICAL TRIAL: NCT06044246
Title: Influence of Human Platelet Derivatives on Dental Implant Osseointegration
Brief Title: Influence of Human Platelet Derivatives on Dental Implant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Afya Sahib Diab Al-radha, Assistant Professor, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUOSU-202103
Record Dates: First submitted 2022-11-24; First posted 2023-09-21 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Platelet-Rich Fibrin; Dental Implantation; Bone Substitute
Keywords: Dental implant; PRF; membrane; osseointegration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Placing dental implant with PRF membrane treatment alone or combined with bone substitute.
  Interventions: Biological: PRF membrane
- control group (No Intervention): Placing dental implant

INTERVENTIONS:
Biological: PRF membrane — Placing implant with PRF membrane treatment
  Arms: experimental group

SUMMARY:
The goal of this randomized controlled trial is to evaluate the benefit of PRF membrane on bone around dental implant in patients who need treatment with dental implant.

Aims of the study:

* To study the effect of PRF membrane (with or without bone substitute on increasing bone dimension around dental implant.
* To investigate the effects of compositions of PRF (platelets count, WBC count) on bone healing.

DETAILED DESCRIPTION:
Materials and methods:

PRF will be obtained from a blood sample that is taken from the patient at the time of surgery in 10-mL tubes, the blood-containing tube is placed in a centrifuge at specially controlled rotations, temperature and time. The result is the separation of blood, basically from two by-products, including PRF. The PRF clot will be placed in specific box ( P.R.F -System; Surgident, CE ) to create a PRF membrane with specific thickness that will be placed on the bone around dental implant.

Evaluation of the results

* Alveolar bone width around dental implant will be measured.
* Histological examination of the tissue that excised during dental implant uncover surgery.
* Evaluate pain by visual analogue score (VAS).
* Estimate the count of WBC and platelets in whole blood will be obtained from a laboratory results.

ELIGIBILITY:
IInclusion criteria

* Non- smoker.
* No medical history of any systemic diseases that affect the bone metabolism.
* Did not receive any systemic drugs.
* Has edentulous area that needs dental implant.

The exclusion criteria were as follows:

* Systemic disease or medication compromising bone and soft tissue healing.
* Pathology in the edentulous region.
* Bruxism.
* Disease of the oral mucosa.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Osseointegration | Immediately after surgery, after 12 weeks (during uncover implant surgery)
  Evaluation of the changes in the degree of osseointegration will be performed using Osstell devise. [Osstell ISQ device. (Stampgatan, Gteborg, Sweden)] The Unit of measurement: ISQ (Implant Stability Quotient), which is a scale from 1 to 100.
Bone width | Baseline (pre-surgery), immediately after the surgery, after 4 weeks, 6 weeks, 8weeks, 10 weeks, and 12 weeks.
  Measure the dimensional changes using special caliper (vernier) measurement tool, to evaluate the changes of bone width around dental implant. the Unit of measurement: millimeter (mm) (Bone and mucosa)

CONTACTS AND LOCATIONS:
Overall Officials: Assis. Prof. Dr. Afya SD Al-radha, Principal Investigator — College of Dentistry, Mustansiriyah University.
Locations (1):
- Kadhimiya Teaching HospitalKadhimiya Educational Hospital, Baghdad, Alkadhmiya City, Iraq

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: following publication. No end date.
Access Criteria: Anyone who wishes to access the data.
URL: https://myaccount.google.com/?utm_source=OGB&utm_medium=app&pli=1

DOCUMENTS (1):
  • Informed Consent Form (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT06044246/ICF_000.pdf